CLINICAL TRIAL: NCT04640545
Title: A Phase I Multi-center Study to Evaluate the Safety ,Tolerability and Efficacy of LBL-007 Combined With Toripalimab or LBL-007 Combined With Toripalimab and Axitinib Tablets in the Treatment of Unresectable or Metastatic Melanoma
Brief Title: A Study to Assess LBL-007 in Combination With Toripalimab and Axitinib Tablets Subjects With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-007-CN-002
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-12

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — toripalimab; Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-007+Toripalimab+Axitinib Tablets (Experimental): Study Part A： LBL-007 +Toripalimab
  Study Part B： LBL-007 +Toripalimab +Axitinib Tablets
  Interventions: Drug: LBL-007; Drug: Toripalimab; Drug: Axitinib Tablets

INTERVENTIONS:
Drug: LBL-007 — LBL-007 will be administered intravenously every two weeks (Q2W) .
Drug: Toripalimab — Toripalimab Injection will be administered by intravenously (Q2W) .
Drug: Axitinib Tablets — Axitinib Tablets On-demand administration

SUMMARY:
A phase I clinical study evaluating LBL-007 in the treatment of subjects with advanced solid tumors

DETAILED DESCRIPTION:
This trial is a multi-center, single-arm, open-label, dose-escalation and expansion phase I study of LBL-007 combined with Toripalimab and Axitinib in the treatment of unresectable or metastatic melanoma.

It is divided into Study Part A and Study Part B. The safety, tolerability, kinetic characteristics, immunogenicity and preliminary efficacy of the subjects were evaluated. Both study part A and study part B are studied in two phases: dose escalation and dose expansion

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent and follow the study treatment plan and visit plan;
2. Aged ≥ 18 years at time of signing informed consent, male or female;
3. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1;
4. Have life expectancy of at least 12 weeks ;
5. Subject with at least one measurable tumor lesion,according to the evaluation standard of solid tumor efficacy (RECIST 1.1).

Exclusion criteria:

1. Subjects are allergic to LBL-007, PD-1 and similar compounds or any component in the prescription;
2. Subjects with active central nervous system metastases (regardless of whether they have received treatment), including symptomatic brain metastases, meningeal metastases, or spinal cord compression, but asymptomatic brain metastases (no progression and/or at least 4 weeks after radiotherapy) No neurological symptoms or signs after surgical resection, and dexamethasone or mannitol treatment is not required);
3. Have received major surgery within 4 weeks before the first administration;
4. Subjects can not tolerate intravenous administration and have difficulty in venous blood collection (if there is a history of fainting needles and bleeding);
5. Women during pregnancy or lactation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Number of subjcects with adverse events and serious adverse events | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  The safety profile of LBL-007 and Toripalimab will be assessed by monitoring the adverse event(AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE)v5.0
Maximum tolerated dose (MTD) | During the first two Cycles(each cycle is 14 days)
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first two cycles.
Dose-limiting toxicities (DLT) | During the first two Cycles(each cycle is 14 days)
  DLT is defined as a toxicities(adverse event at least possibly related to LBL-007 and Toripalimab )occurring during the DLT observation period(the initial 28 days).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Defined as the percentage of subjects having a Complete Response or Partial Response(ORR, including after immunotherapy complete response (iCR) and partial response (iPR)),will be determined by investigator assessment of radiographic disease assessments per RECIST v1.1. and iRECIST.
Duration of Response(DOR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Defined as the time from earliest date of disease response (CR 、PR、iCR、iPR) until earliest date of disease progression, as determined by investigator assessment of radiographic disease per RECIST v1.1 and iRECIST, or death from any cause, if occurring sooner than progression.
Disease Control Rate(DCR) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Defined as percentage of participants having CR, PR, iCR，iPR or SD as best on-study response
Steady state Area under the serum concentration versus time curve（AUCss） | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  To determine the PK profile of LBL-007 in combination with Toripalimab
Steady state Maximum serum concentration (Cmax,ss) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  To determine the PK profile of LBL-007 in combination with Toripalimab
Steady state Time to reach maximum serum concentration (Tmax,ss) | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  To determine the PK profile of LBL-007 in combination with Toripalimab
Pharmacodynamic (PD) index | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  The PD evaluation index is the LAG-3 receptor occupancy rate in peripheral blood
Immunogenicity index | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal (28+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity evaluation indicators are the incidence of anti-drug antibodies (ADA) and the incidence of neutralizing antibodies (if applicable) in the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Prof, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - the First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No